CLINICAL TRIAL: NCT02314104
Title: Analgesic Efficacy of Transversus Abdominis Plane Block Versus Local Injection in Postoperative Pain Management Following Minimally Invasive Gynecological Surgery
Brief Title: Efficacy of Transversus Abdominis Plane Block Versus Local Injection of Pain Medication
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Liberman, Eric, D.O. (Individual)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 11-02
Record Dates: First submitted 2014-12-08; First posted 2014-12-10 (Estimated); Results first posted 2015-04-14 (Estimated); Last update posted 2015-04-14 (Estimated); Status verified 2015-04

CONDITIONS: Pain, Postoperative
Keywords: Surgical procedures, Minimally invasive; Nerve block; Anesthetics, Local
MeSH Terms: conditions — Pain, Postoperative | interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Treatment TAP, placebo local injection (Active Comparator): Treatment TAP block was 30 mL 0.5% ropivacaine bilaterally. Placebo local injection was 2 mL of 0.9% normal saline at each port site.
  Interventions: Drug: ropivacaine
- Placebo TAP, treatment local injection (Active Comparator): Placebo TAP was 30 mL of 0.9% normal saline bilaterally. Treatment local injection was 2 mL of 0.5% ropivacaine at each port site.
  Interventions: Drug: ropivacaine
- Treatment TAP, treatment local injection (Active Comparator): Treatment TAP was 30 mL of 0.5% ropivacaine bilaterally. Treatment local injection was 2 mL of 0.5% ropivacaine at each port site.
  Interventions: Drug: ropivacaine

INTERVENTIONS:
Drug: ropivacaine — Treatment local injection was 2 mL of 0.5% ropivacaine at each port site. Treatment TAP was 30 mL of 0.5% ropivacaine bilaterally.
  Other Names: Naropin

SUMMARY:
The purpose of this study is to determine if there is a better method of administering pain medication prior to minimally invasive gynecological surgery so that postoperative pain and/or narcotic usage may be minimized. Currently, no standard of care exists regarding the use of local pain medications in minimally invasive gynecological surgery and practices vary widely among physicians, even within the same institution.

The two methods of preemptive pain medication that this study will be looking at is the transversus abdominis plane (TAP) block and the local injection of pain medication at the areas of the skin incisions. TAP block is a procedure performed by a specially trained pain management anesthesiologist in which there is an injection of a local pain medication into the abdominal wall, specifically in a space where the nerves that are responsible for postoperative pain reside. This procedure blocks the ability of the nerves to sense pain and has been found to be successful in decreasing postoperative pain in a number of procedures. The local injection of pain medications at the incision sites has also been found to be beneficial in decreasing postoperative pain. However, it is not known whether one method is superior to the other in decreasing postoperative pain or if the combination of both is best.

Patients that chose to participate are randomly (by chance) assigned to one of three groups: 1) TAP block with pain medication and local injection of normal saline (water) at the incision sites 2) TAP block with normal saline and local injection of pain medication at the incision sites or 3) TAP block with pain medication and local injection of pain medication at the port sites. These procedures are performed while the patient is asleep. Patients will be asked to record their level of pain on a standardized pain scale at one hour, six hours, and twenty-four hours after the surgery. All patients are provided with standard postoperative pain medications as needed.

The hypothesis is that patients receiving both TAP block and local injection of pain medication at the port sites will have less pain postoperatively and require a smaller amount of narcotics than those that receive either the TAP block or local injection of pain medication alone.

DETAILED DESCRIPTION:
This is a prospective, single center, double-blinded, multi-arm parallel group study conducted at a university affiliated medical center. Study approval was obtained from the Saint Barnabas Medical Center institutional review board, and written informed consent was obtained from all study participants.

Patients were randomly assigned to one of three parallel groups in a 1:1:1 ratio, to receive either: treatment transversus abdominis plane (TAP) block and placebo local injection, placebo TAP block and treatment local injection, or treatment TAP block and treatment local injection. This study took place at Saint Barnabas Medical Center in Livingston, New Jersey from May 2011 to October 2013. Patients were recruited from the offices of ten different gynecological surgeons in private practice. Two of the surgeons were gynecological oncologists, and the remainder were general obstetricians/gynecologists that perform minimally invasive gynecological surgery. The TAP blocks were administered by one of four anesthesiologists.

Patients were consented and enrolled in the study by blinded obstetrical and gynecological residents while the patients were in the preoperative area. Each patient was given a standardized informed consent packet detailing the study. Once a patient gave informed consent and was enrolled in the study, independent pharmacists were notified of their enrollment. The pharmacists then assigned participants to one of three possible interventions based on a computer-generated randomization list that was created by the principal investigator prior to commencement of patient enrollment. The pharmacist assigned patients into their appropriate intervention based upon what number participant the patient was in the study. The pharmacist then dispensed the study medications into identical 30 mL syringes labeled study drug and placed them in brown paper bags. The study medication to be administered via TAP block was placed in two 30 mL syringes and placed in a brown paper bag. The study medication to be used for local injection was placed in a single 30 mL syringe and placed in a separate brown paper bag. These bags were then brought to the operating room where they were to be administered. The bag containing the two syringes was given to the anesthesiologists performing the TAP block and the bag with the single syringe was handed to the scrub tech that then later distributed it to the surgeons. The patients, all healthcare providers, and data collectors were blinded as to group allocation. Additionally, both ropivacaine and normal saline are clear and indistinguishable from one another.

The interventions were administered in the operating room once the patients had been placed under general anesthesia, prior to skin incisions. The TAP blocks were administered under ultrasound guidance.

Patients were then prepped and draped for surgery. Prior to proceeding to skin incisions the surgeons administered 2 mL of local injection subcutaneously at the intended port site locations. If additional port sites were deemed necessary during the procedure study drug was administered in a similar fashion prior to those skin incisions being made.

Postoperatively all patients received a standardized analgesia regimen. Specifically, for mild pain, oxycodone/acetaminophen 5/325 mg one tablet orally every four hours; for moderate pain, oxycodone/acetaminophen 5/325 mg two tablets orally every six hours, and for severe pain, hydromorphone 1 mg every 3 hours intravenously.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Undergoing gynecological robotic and/or laparoscopic surgery
* Overnight hospitalization expected

Exclusion Criteria:

* Fibromyalgia
* Chronic pelvic pain
* Relevant drug allergy
* Conversion to laparotomy
* Pregnant

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2011-05; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric C Liberman, D.O., Principal Investigator — St. Barnabas Medical Center; Thad Denehy, M.D., Principal Investigator — St. Barnabas Medical Center
Locations (1):
- Saint Barnabas Medical Center, Livingston, New Jersey, United States

REFERENCES:
- [Background] Carney J, McDonnell JG, Ochana A, Bhinder R, Laffey JG. The transversus abdominis plane block provides effective postoperative analgesia in patients undergoing total abdominal hysterectomy. Anesth Analg. 2008 Dec;107(6):2056-60. doi: 10.1213/ane.0b013e3181871313. PMID 19020158
- [Background] El Hachem L, Small E, Chung P, Moshier EL, Friedman K, Fenske SS, Gretz HF 3rd. Randomized controlled double-blind trial of transversus abdominis plane block versus trocar site infiltration in gynecologic laparoscopy. Am J Obstet Gynecol. 2015 Feb;212(2):182.e1-9. doi: 10.1016/j.ajog.2014.07.049. Epub 2014 Aug 1. PMID 25088860
- [Background] Hebbard P, Fujiwara Y, Shibata Y, Royse C. Ultrasound-guided transversus abdominis plane (TAP) block. Anaesth Intensive Care. 2007 Aug;35(4):616-7. No abstract available. PMID 18020088
- [Background] Kane SM, Garcia-Tomas V, Alejandro-Rodriguez M, Astley B, Pollard RR. Randomized trial of transversus abdominis plane block at total laparoscopic hysterectomy: effect of regional analgesia on quality of recovery. Am J Obstet Gynecol. 2012 Nov;207(5):419.e1-5. doi: 10.1016/j.ajog.2012.06.052. Epub 2012 Jun 29. PMID 22840413
- [Background] Rafi AN. Abdominal field block: a new approach via the lumbar triangle. Anaesthesia. 2001 Oct;56(10):1024-6. doi: 10.1046/j.1365-2044.2001.02279-40.x. No abstract available. PMID 11576144

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment TAP, Placebo Local Injection | Placebo TAP, Treatment Local Injection | Treatment TAP, Treatment Local Injection
Started | 71 | 78 | 71
Completed | 57 | 58 | 53
Not Completed | 14 | 20 | 18

BASELINE CHARACTERISTICS:
Population: arm 1: 6 baseline data lost, 3 did not report scores, 1 surgery cancelled after TAP, arm 2: 6 did not report scores, 6 baseline data lost, 1 developed allergy, 1 TAP given after surgery, 1 never received TAP arm 3: 6 did not report scores, 2 developed allergy, 2 surgery cancelled after TAP, 1 re-operated, 1 discharged immediately
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment TAP, Placebo Local Injection | Placebo TAP, Treatment Local Injection | Treatment TAP, Treatment Local Injection | Total
Number analyzed (Participants) | 61 | 63 | 59 | 183
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.8 (11.3) | 52.0 (9.9) | 56.1 (11.0) | 54.0 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61 | 63 | 59 | 183
  Male | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 61 | 63 | 59 | 183
BMI (m/kg2) [Mean (Standard Deviation); unit: kg/m^2] | 30.5 (7.4) | 31.9 (7.0) | 29.9 (7.5) | 30.8 (7.3)
Weight (kg) [Mean (Standard Deviation); unit: kg] | 80.8 (20.5) | 85.9 (18.4) | 79.2 (20.0) | 82.0 (19.6)
Height (inches) [Mean (Standard Deviation); unit: inches] | 64 (2.6) | 64.7 (2.5) | 64.1 (2.5) | 64.3 (2.5)

OUTCOME MEASURES:

1. Primary Outcome: Postoperative Pain on a Visual Analogue Pain Scale at One Hour Postoperatively
Description: A Visual Analogue Scale was used. The scale range was 0 to 10 in increments of one. 0 was no pain and 10 was worst pain possible.
Time Frame: one hour postoperatively
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment TAP, Placebo Local Injection | Placebo TAP, Treatment Local Injection | Treatment TAP, Treatment Local Injection
Number analyzed (Participants) | 57 | 58 | 53
units on a scale | 4.04 (2.9) | 5.09 (2.46) | 4.4 (2.53)

2. Primary Outcome: Postoperative Pain on a Visual Analogue Pain Scale at Six Hours Postoperatively
Description: as for outcome 1
Time Frame: six hours postoperatively
Population: Arm 2: 6 hour pain score not obtained on one subject Arm 3: 6 hour pain score not obtained on one subject
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment TAP, Placebo Local Injection | Placebo TAP, Treatment Local Injection | Treatment TAP, Treatment Local Injection
Number analyzed (Participants) | 57 | 57 | 52
units on a scale | 3.53 (2.62) | 3.5 (1.93) | 3.33 (2.53)

3. Primary Outcome: Postoperative Pain on a Visual Analogue Pain Scale at Twenty-four Hours Postoperatively
Description: as for outcome 1
Time Frame: twenty-four hours postoperatively
Population: Arm 1: one subject discharged prior to obtaining 24 hour pain score Arm 2: one subject discharged prior to obtaining 24 hour pain score Arm 3: four subjects discharged prior to obtaining 24 hour pain score
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment TAP, Placebo Local Injection | Placebo TAP, Treatment Local Injection | Treatment TAP, Treatment Local Injection
Number analyzed (Participants) | 56 | 57 | 49
units on a scale | 3.36 (2.15) | 3.56 (2.13) | 3.51 (2.59)

4. Secondary Outcome: Time Until First Request for Pain Medication
Time Frame: up to twenty-four hours postoperatively
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Treatment TAP, Placebo Local Injection | Placebo TAP, Treatment Local Injection | Treatment TAP, Treatment Local Injection
Number analyzed (Participants) | 57 | 58 | 53
minutes | 46 [18 to 104] | 31 [20 to 56] | 28 [13 to 78]

5. Secondary Outcome: Total Narcotic Usage in Morphine Equivalents
Time Frame: up to twenty-four hours postoperatively
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Treatment TAP, Placebo Local Injection | Placebo TAP, Treatment Local Injection | Treatment TAP, Treatment Local Injection
Number analyzed (Participants) | 57 | 58 | 53
mg | 20.09 (11.6) | 23.14 (12.3) | 20.68 (12.8)

ADVERSE EVENTS:
Arm/Group | Treatment TAP, Placebo Local Injection | Placebo TAP, Treatment Local Injection | Treatment TAP, Treatment Local Injection
Serious Adverse Events (participants affected / at risk) | 0/71 | 0/78 | 0/71
Other Adverse Events (participants affected / at risk) | 0/71 | 0/78 | 0/71

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes